CLINICAL TRIAL: NCT04196842
Title: Heart Failure Precision Medicine Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1471560
Record Dates: First submitted 2019-11-12; First posted 2019-12-12 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Heart Failure
Keywords: Heart Failure; Multi-omics; Phenomapping; Precision medicine; Telemonitoring
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinded until intervention is assigned to subject
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemonitoring (Experimental): Blood pressure and heart rate monitoring, scale, activity tracker.
  Interventions: Device: Telemonitoring devices
- No intervention (No Intervention): No intervention.

INTERVENTIONS:
Device: Telemonitoring devices — Set of telemonitoring devices: heart rate and blood pressure monitor, scale and activity tracker.
  Arms: Telemonitoring

SUMMARY:
The study aims to test the hypothesis that multi-omics studies can identify Heart Failure profiles at risk of adverse outcomes and evaluate a telemonitoring intervention in the optimization of guideline-directed medical therapy.

DETAILED DESCRIPTION:
In the US, the estimated prevalence of Heart Failure (HF) is 6.2 million and increasing. The mortality approaches 50% within 5 years of diagnosis and HF is the main cause of hospitalization among patients over 65 years of age. Information on molecular states may enhance understanding of causes and pathophysiological processes, improve risk prediction, identify new therapeutic targets, and improve subclassification for targeted therapy. Time-dependent phenomapping has been used to identify clinical and genomic differences in a longitudinal fashion, which provides a mechanistic link underlying pathophysiology of the disease and associated outcomes. Studies including high-throughput molecular approaches (multi-omics) along with time-dependent phenomapping would likely be even more powerful. The overarching hypothesis of the study is that the integration of Multi-Omics studies with clinical variables can be implemented to identify patients at risk of adverse outcomes. To test this hypothesis we propose: (1) Longitudinal profiling based on clinical data; (2) Longitudinal Multi-Omics Profiling; and (3) randomized of a telemonitoring intervention (Sensor Profiling) and the effectiveness in the optimization of guideline-directed medical therapy. To achieve these aims we propose to: (1) recruit a cohort of 1000 participants; (2) perform cardiovascular clinical characterization from electronic medical records; (3) perform multi-omics studies and (4) randomization of a telemonitoring intervention in the optimization of guideline-directed medical therapy. Proving these hypotheses would identify different meaningful clinical groups of patients within a cohort of patients with similar clinical conditions, health care providers would have a better understanding of the heterogeneity of the disease and the need for different preventive and therapeutic approaches in the context of precision medicine.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Heart failure
* Objective evidence of cardiac abnormality of structure or function (abnormal ECHO) or elevated levels of B-type natriuretic peptide (>100 pg/ml)
* HF stage B-D and class I-IV

Exclusion Criteria:

* Patients unable to consent
* Inability to comply with the protocol and follow-up requirements
* Patients unable to use a smartphone
* Patients assessed irregularly (less than two visits in one year)
* History of HTx
* Use of Mechanical circulatory support device (MCSD)
* Comorbidities that, according to the PI, have the potential to interfere with the interpretation of the results

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-16 (Actual); Primary Completion 2026-10-16 (Estimated); Study Completion 2026-10-16 (Estimated)

PRIMARY OUTCOMES:
Rate of adverse outcomes in heart failure | Five years from enrollment
  Rate of Mortality (all cause), hospitalization, Mechanical circulatory support device (MCSD) or heart transplant (HTx)

SECONDARY OUTCOMES:
Disease progression | Five years from enrollment
  Disease severity (ACC/AHA Heart Failure classification system)

OTHER OUTCOMES:
Percentage of guideline-directed medical therapy (GDMT). | One year from enrollment
  Percentage of GDMT target doses

CONTACTS AND LOCATIONS:
Overall Officials: Martin Cadeiras, MD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/study-of-using-omics-genes-metabolites-and-proteins-from-blood-and-heart-tissue-to-learn-more-about-heart-disease-124030/